CLINICAL TRIAL: NCT04792775
Title: PTSD Treatment and Emotion Regulation Skills Training for Veterans With Military Sexual Trauma
Brief Title: PTSD Treatment and Emotion Regulation Skills Training for Veterans With Military Sexual Trauma (PE+ER)
Acronym: PE+ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00107912
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Stress Disorders, Post-Traumatic; Anxiety Disorders; Mental Disorder; Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Mental Disorders; Stress Disorders, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prolonged Exposure + Emotion Regulation Skills Training (Experimental): Twelve, 90-minute sessions of Prolonged Exposure (PE) with Dialectical Behavior Therapy (DBT) Emotion Regulation Skills Training.
  Interventions: Behavioral: PE+ER

INTERVENTIONS:
Behavioral: PE+ER — PE includes the following components: a) psychoeducation about the common reactions to traumatic events and presentation of the treatment rationale b) repeated in vivo exposure to traumatic stimuli, c) repeated, prolonged, imaginal exposure to traumatic memories, and d) relapse prevention strategies and further treatment planning (session 12). DBT Emotion Regulation Skills is integrated as part of this intervention. DBT training provides skills to understand, name, experience and tolerate emotions, as well as skills to change negative emotional responses and to reduce vulnerability to emotion dysregulation (Linehan et al., 2015). The current project includes an adapted 3- session individual emotion regulation skills training intervention to be implemented concurrently with PE which consists of initial teaching/instruction and brief skills review for the remainder of PE treatment.

SUMMARY:
Prior research has found that Veterans with military sexual trauma (MST) who have more difficulties with emotion regulation were more likely to drop out of PTSD treatment prematurely. The purpose of this pilot study is to determine whether integrating evidence-based emotion regulation skills training with a scientifically validated treatment for PTSD called Prolonged Exposure (PE), will enhance PTSD treatment retention and 'dose received' and subsequently improve treatment outcomes for MST-related PTSD and difficulties with emotion regulation. Results from this project that examine the feasibility of integrating these two treatments will provide methodological evidence and justification for a randomized control trial, if warranted.

DETAILED DESCRIPTION:
The purpose of this study is to learn ways to improve treatments for women with military sexual trauma (MST). The researchers want to learn whether combining evidence-based emotion regulation skills training with a trauma-focused therapy improves treatment outcomes. An evidence-based trauma treatment known as Prolonged Exposure will be used. Emotion regulation skills will also be included in treatment. Veterans with a positive or sub threshold diagnosis of PTSD who experienced a military sexual trauma (MST) will be included. Participants will complete up to twelve 90 minute sessions of PE with Dialectical Behavior Therapy (DBT) Emotion Regulation Skills Training followed by a post-treatment assessment. All aspects of the project including consent, baseline, treatment and follow-up will be completed either in person or via videoconferencing. Fifteen participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* MST-related index event
* Diagnosis of PTSD related to MST assigned on the basis of the Clinician Administered PTSD Scale (CAPS; Weathers et al., 2013)
* Difficulties with emotion regulation as identified by the Difficulties with Emotion Regulation Scale (DERS; Gratz & Roemer, 2004; although there is no clinical cutoff for the DERS, a total score of 99 is indicative of one standard deviation above average difficulties with emotion regulation for women).

Exclusion Criteria:

* Having a household member who is already enrolled in the study
* Active psychosis or dementia at screening
* Suicidal ideation with clear intent
* Current moderate to severe Substance Use Disorder
* Concurrent enrollment in a clinical trial for PTSD or depression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-01-19 (Actual)

PRIMARY OUTCOMES:
Clinical Administrated PTSD Scale (CAPS) | 13 weeks
  The Clinician Administered PTSD (Posttraumatic stress disorder) Scale (CAPS) is a 30-item structured interview that corresponds to the Diagnostic and Statistical Manual of Mental Disorders, 5th Version (DSM-V) criteria for PTSD. The CAPS can be used to make a current (past month) or lifetime diagnosis of PTSD or to assesses symptoms over the past week. CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). A symptom cluster score may also be calculated for dissociation by summing items 19 and 20. Scores range from 0 to 80.

SECONDARY OUTCOMES:
PTSD Checklist, 5th Version (PCL-5) | 13 weeks
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD, and making a provisional PTSD diagnosis. Description information provided by the National Center for PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Muzzy, MRA, MLIS, Principal Investigator — Medical University of South Carolina; Amanda Gilmore, PhD, Principal Investigator — Georgia State University
Locations (1):
- Ralph H. Johnson VAMC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No